CLINICAL TRIAL: NCT02764593
Title: Safety Evaluations of Nivolumab (Anti-PD-1) Added To Chemotherapy (CRT) Platforms In Patients With Intermediate And High-Risk Local-Regionally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Safety Testing of Adding Nivolumab to Chemotherapy in Patients With Intermediate and High-Risk Local-Regionally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RTOG Foundation, Inc. (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 3504; RF 3504 (Other: RTOG Foundation); CA209-410 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: Head and Neck Squamous Cell Carcinoma; HNSCC; Nivolumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Cisplatin; Cetuximab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Nivolumab + Cisplatin) (Experimental): Patients will receive Nivolumab via IV administration every 14 days for 10 doses starting 14 days prior to IMRT. Cisplatin will be given weekly. IMRT will be given at 5 fractions per week for 7 weeks for a dose of 70 Gy. Adjuvant nivolumab every 28 days for 7 doses will be administered starting 3 months after end of chemoradiation. Adjuvant administration of nivolumab may be discontinued if more than 4 of first 8 patients receive less than 7 doses.
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Radiation: IMRT
- Arm 2 (Nivolumab + High-dose Cisplatin) (Experimental): Patients will receive Nivolumab via IV administration starting 14 days prior to IMRT, then Day 1 of IMRT and then every 21 days for 6 doses. Cisplatin will be given every 21 days for 3 doses. IMRT will be given at 5 fractions per week for 7 weeks for a dose of 70 Gy. Adjuvant nivolumab every 28 days for 7 doses will be administered starting 3 months after end of chemoradiation. Adjuvant administration of nivolumab may be discontinued if more than 4 of first 8 patients receive less than 7 doses.
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Radiation: IMRT
- Arm 3 (Nivolumab + Cetuximab) (Experimental): Patients will receive Nivolumab via IV administration every 14 days for 10 doses starting 14 days prior to IMRT. Cetuximab will be given for 7 doses. IMRT will be given at 5 fractions per week for 7 weeks for a dose of 70 Gy. Adjuvant nivolumab every 28 days for 7 doses will be administered starting 3 months after end of chemoradiation. Adjuvant administration of nivolumab may be discontinued if more than 4 of first 8 patients receive less than 7 doses.
  Interventions: Drug: Nivolumab; Drug: Cetuximab; Radiation: IMRT
- Arm 4 (Nivolumab + IMRT) (Experimental): Patients will receive Nivolumab via IV administration every 14 days for 10 doses starting 14 days prior to IMRT. IMRT will be given at 5 fractions per week for 7 weeks for a dose of 70 Gy. Adjuvant nivolumab every 28 days for 7 doses will be administered starting 3 months after end of chemoradiation. Adjuvant administration of nivolumab may be discontinued if more than 4 of first 8 patients receive less than 7 doses.
  Interventions: Drug: Nivolumab; Radiation: IMRT

INTERVENTIONS:
Drug: Nivolumab — Anti-PD-1 targeted immunotherapy
  Other Names: Opdivo
Drug: Cisplatin — Anti-cancer alkylating agent
  Other Names: Platinol
  Arms: Arm 1 (Nivolumab + Cisplatin); Arm 2 (Nivolumab + High-dose Cisplatin)
Drug: Cetuximab — Epidermal Growth Factor Receptor (EGFR) antagonist
  Other Names: Erbitux
  Arms: Arm 3 (Nivolumab + Cetuximab)
Radiation: IMRT — High-precision radiotherapy
  Other Names: Intensity Modulated Radiation Therapy

SUMMARY:
This study will evaluate the safety of adding nivolumab to several chemotherapy platforms with weekly cisplatin, high-dose cisplatin, cetuximab or radiation therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed diagnosis of HNSCC of the oral cavity, oropharynx, larynx, or hypopharynx.
* Intermediate-risk group: Oropharynx cancer that is p16-positive by immunohistochemistry with smoking status > 10 Pack-years, stage T1-2N2b-N3 OR ≤ 10 pack-years, stage T4N0-N3 or T1-3N3.
* High-risk group: Oral cavity, larynx, hypopharynx, or p16-negative oropharynx cancer, stage T1-2N2a-N3 or T3-4-N0-3 based on the following diagnostic workup:

  * Mandatory submission of H&E and p16 stained slides for central review of p16 staining is required for oropharyngeal patients and H&E stained slide block (or punch biopsy of paraffin block) for PD-L1 expression analysis for all patients
  * History/physical examination within 28 days prior to registration
  * Examination by Radiation Oncologist, Medical Oncologist, and Ear, Nose, Throat (ENT) or Head & Neck Surgeon within 28 days prior to registration
  * Fiberoptic exam with laryngopharyngoscopy within 28 days prior to registration
  * Diagnostic quality, cross sectional imaging of the thorax within 28 days prior to registration; 18-F-FDG-PET/CT or conventional CT are acceptable.
  * Diagnostic quality CT or MRI of neck, with contrast, within 28 days prior to registration; a 18-F-FDG-PET/CT of the neck only is acceptable as a substitute if the CT is of diagnostic quality and with IV contrast.
* Age ≥ 18 years
* The trial is open to both genders

Exclusion Criteria:

* Definitive clinical or radiologic evidence of distant (beyond cervical lymph node and neck tissue) metastatic disease.
* Patients with oral cavity cancer are excluded from participation if resection of the primary tumor is considered technically feasible by an oral or head and neck cancers surgical subspecialist.
* Carcinoma of the neck of unknown primary site origin (even if p16-positive).
* Absence of RECIST, v. 1.1 defined measurable disease.
* Gross total excision of both primary and nodal disease; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease. Patients with RECIST, v. 1.1 evaluable remaining cancer either in the neck or primary site remain eligible.
* Simultaneous primary cancers or separate bilateral primary tumor sites.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
* Prior systemic chemotherapy for the study cancer.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* Patients with active autoimmune disease, with exceptions of vitiligo, type I diabetes mellitus, hypothyroidism and psoriasis.
* Use of systemic corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration, with exception of inhaled or topical steroids.
* Known immunosuppressive disease, for example HIV infection or history of bone marrow transplant or chronic lymphocytic leukemia (CLL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06; Primary Completion 2018-09-25 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | From the first dose of nivolumab to 28 days after the completion of radiation therapy.
  A nivolumab attributable, dose-limiting toxicity (DLT) will be defined as follows:
  1) Any ≥ grade 3 adverse event (CTCAE, v. 4) that is related to nivolumab that does not resolve to grade 1 or less within 28 days; 2) A delay in radiotherapy of > 2 weeks due to toxicity related to nivolumab; 3) Inability to complete radiotherapy due to toxicity related to nivolumab; 4) Inability to receive an adequate dose (≥ 70%) of cisplatin (Arm 1 and 2) or cetuximab (Arm 3) due to toxicity definitely related to nivolumab.

CONTACTS AND LOCATIONS:
Overall Officials: Maura Gillison, MD, PhD, Principal Investigator — RTOG Foundation; Robert Ferris, MD, PhD, Principal Investigator — RTOG Foundation
Locations (11):
- United States (11):
  - Stanford Cancer Institute, Palo Alto, California
  - University of Florida Cancer Center at Orlando Health, Orlando, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - UPMC - Shadyside Hospital, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gillison ML, Ferris RL, Harris J, Colevas AD, Mell LK, Kong C, Jordan RC, Moore KL, Truong MT, Kirsch C, Chakravarti A, Blakaj DM, Clump DA, Ohr JP, Deeken JF, Gensheimer MF, Saba NF, Dorth JA, Rosenthal DI, Leidner RS, Kimple RJ, Machtay M, Curran WJ Jr, Torres-Saavedra P, Le QT. Safety of Nivolumab Added to Chemoradiation Therapy Platforms for Intermediate and High-Risk Locoregionally Advanced Head and Neck Squamous Cell Carcinoma: RTOG Foundation 3504. Int J Radiat Oncol Biol Phys. 2023 Mar 15;115(4):847-860. doi: 10.1016/j.ijrobp.2022.10.008. Epub 2022 Oct 11. PMID 36228746

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT02764593/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT02764593/ICF_001.pdf